CLINICAL TRIAL: NCT03721432
Title: The Effect of Oral Pregabalin on Epidural-induced Shivering and Epidural Characteristics in Gynecological Surgeries, a Prospective Randomized Double-blind Study
Brief Title: The Effect of Oral Pregabalin on Epidural-induced Shivering and Epidural Characteristics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Tarel Al Menisy, Associate professor, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FM-BSU REC 006/2018
Record Dates: First submitted 2018-10-10; First posted 2018-10-26 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Epidural Anesthesia; Shivering
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: sealed opaque numbered envelopes indicating the group of each patient, carried out by an independent anesthesiologist and given to the ward nurse
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pregabalin group (P) (Experimental): received pregabalin 150 mg capsules (Lyrica®,Pfizer) sixty minutes prior to the epidural insertion.
  Interventions: Drug: Pregabalin 150mg
- Control group (C) (Placebo Comparator): received placebo capsules sixty minutes prior to epidural insertion.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Pregabalin 150mg — pregabalin 150 mg capsules (Lyrica®,Pfizer) given 60 minutes prior to epidural anesthesia
  Other Names: Lyrica
  Arms: Pregabalin group (P)
Drug: Placebo oral capsule — Placebo oral capsule given 60 minutes prior to epidural anesthesia
  Arms: Control group (C)

SUMMARY:
* Background: The previous reports tried to reduce shivering and improve neuroaxial anesthesia characteristics by the systemic use of different drugs. This study was directed to evaluate the effect of pregabalin premedication on both shivering and epidural outcome data following single shot loading.
* Patients and Methods: Eighty patients, ASA grade I and II, undergoing surgeries under epidural anesthesia were studied. The patients were divided into two groups: Pregabalin group and Control group in which the patients received 150 mg of pregabalin and placebo capsules respectively sixty minutes prior to surgery. Following epidural loading, the onset and degree of shivering were compared between the two groups. Also, the epidural outcome including onset, level and duration were traced and compared. The perioperative hemodynamics, sedation scores, patient satisfaction and side effects were followed up and registered.

DETAILED DESCRIPTION:
After obtaining the ethical committee approval of Beni Suef University hospital, in Egypt and an informed consent from the patients, Eighty female patients with an American society of Anesthegiologists physical status (ASA) I-II who were undergoing gynecological surgery (Posterior repair and transobturator transfixation) under epidural anesthesia, were enrolled in this randomized double -blind study in May 2018.

The patients were excluded from the study if ASA class was more than II, anticipated difficult epidural insertion or there was any contraindication to epidural anesthesia, if any patient developed wet or bloody tab, or the patients were under psychotropic or antiepileptic therapy.

The 80 Patients were randomly allocated into one of two groups (using sealed opaque numbered envelopes indicating the group of each patient, carried out by an independent anesthesiologist and given to the ward nurse) [40 patients in each group]:

* Pregabalin group (P), [n=40]: received pregabalin 150 mg capsules (Lyrica®,Pfizer) sixty minutes prior to the epidural insertion.
* Control group (C), [n=40]: received placebo capsules sixty minutes prior to epidural insertion.

Prior to administration of study drugs, mean arterial blood pressure (MAP), heart rate (HR), oxygen saturation (SpO2), and tympanic temperature (T temp) were taken as [baseline reading]. Upon reaching the operation theater, a second set of readings were taken [preoperative reading], together with sedation score using a 4 points "Modified Wilson" Sedation Scale [1=awake; 2=drowsy but arousable to command; 3= asleep but arousable to mild physical stimulation; and 4= asleep but not arousable to mild physical stimulation].

On the operating table and after attaching the standard monitoring [5 lead ECG, pulse oximetry, non-invasive arterial blood pressure], the epidural anesthesia was standardized for all patients. After intravenous infusion of 500 ml of lactated Ringer's solution in a wide-bore canula, the epidural catheter was inserted in a lateral position. Following the exclusion of both subarachnoid and intravascular insertion of the catheter, a loading epidural dose of 10 ml levo-bupivacaine 0.5% and 50 mcg fentanyl were injected.

The hemodynamic readings [MAP, HR and SpO2] were monitored and registered every 5 minutes (as routine practice) and tympanic temperature [T temp] was taken upon arrival to operating room, after activation of epidural, then every 15 minutes till the end of surgery.

Intraoperatively, arterial blood pressure was maintained within 20 % of the baseline readings using intravenous boluses of Lactated Ringer's solution and 6 mg increments of ephedrine (if required). Bradycardia (HR less than 60 beats per minutes) was treated with intravenous atropine boluses 0.6 mg.

Also, all patients were active warmed using a convection machine (hot air blower).

Shivering (as a primary outcome) was graded by a blinded observer during the intraoperative and postoperative period using the scale validated by Crossley and Mahajan and Tsai and Chu: [0= no shivering, 1= piloerection or peripheral vasoconstriction but no visible shivering, 2= muscular activity in only one muscle group, 3= muscular activity in more than one muscle group but not generalized shivering, 4= shivering involving the whole body]. Grades 3, and 4 shivering for at least 3 minutes were considered positive, and maximum shivering was considered if generalized shivering interfering with ECG monitoring. Positive shivering or lower grade shivering but described as distressful by the patient were treated with intravenous administration of meperidine 20 mg. If no improvement after this management, the patient was excluded from the study.

For the selection of safe and effective anti-shivering treatment, the medications were revised and meperidine in this small dose was picked up due to its effectiveness in treatment and the epidural parameters will not be significantly affected when compared to ketanserine, doxapram, clonidine, magnesium, ketamine, orphenadrine, methylphenidate, pentazocin and nefopam.

At the end of surgery, the patients were transferred to PACU (for one hour), where hemodynamics and tympanic temperature were taking (every 15 minutes). Shivering was also observed and scaled and treated the same way as intraoperatively. Patients were only discharged from PACU if modified Aldrete score was ≥ 9 after registering and treating any other complications.

Postoperatively, when the patients started to experience pain at the surgical site and according to the acute pain management protocol by the anesthesia department in the hospital, a loading of levo-bupivacaine 0.125% 8 ml was given followed by infusion of levo-bupivacaine 0.125% and fentanyl 2mcg/ ml at a rate of 6 ml/hour.

Any perioperative complications (e.g. bradycardia, hypotension, desaturation or nausea and vomiting) were observed, registered and treated appropriately.

The following were observed (by anaesthetist blinded to the studied drugs):

* Demographic data (age, weight and height), duration of surgery (in minutes).
* Tympanic temperature (T temp.) in Celsius degree as baseline (before drug intake), preoperative (on arrival to operating room), after epidural loading, then every 15 minutes intraoperative.
* Shivering (as a primary outcome): incidence of positive shivering (at any time), incidence of maximum shivering (at any time) and median and range of shivering severity between the two studied groups.
* Sedation: assessed 60 minutes after studied drug in take (preoperatively).
* Epidural characteristics (as secondary outcome): onset of the block (the time from epidural loading until feeling of numbness in the lower extremities), duration of the block (the time from the onset till starting feeling of pain at the surgical site) and level of the block (assessed by the ice technique).
* Meperidine consumption: total consumed dose of meperidine in both groups.

ELIGIBILITY:
Inclusion Criteria:

* adults female patients (20 - 60 years old)
* with an American society of Anesthegiologists physical status (ASA) I-II
* undergoing gynecological surgery

Exclusion Criteria:

* ASA class was more than II,
* anticipated difficult epidural insertion
* any contraindication to epidural anesthesia, if any patient developed wet or bloody tab, or the patients were under psychotropic or antiepileptic therapy.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female patients
Enrollment: 77 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
- Shivering | starting from epiural injection, up to 60 minutes after epidural anesthesia
  incidence of positive shivering ,
Shivering | starting from epiural injection, up to 60 minutes after epidural anesthesia
  incidence of maximum shivering

SECONDARY OUTCOMES:
- Epidural characteristics | from epidural injection till numbing sensation (approximately 10 minutes)
  onset of the block (the time from epidural loading until feeling of numbness in the lower extremities)
Epidural characteristics | from epidural onset to starting feeling pain (approximately 90 minutes)
  duration of the block (the time from the onset till starting feeling of pain at the surgical site)

CONTACTS AND LOCATIONS:
Locations (1):
- Beni suef university hospiital, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
participant data are confidential and can only be exposed uopn legal reasons